CLINICAL TRIAL: NCT01364051
Title: Phase I Study of the Combination of the VEGFR Inhibitor, AZD2171, and MEK Inhibitor, AZD6244, in the Treatment of Solid Malignancies
Brief Title: Cediranib Maleate and Selumetinib Sulfate in Treating Patients With Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02906; NCI-2012-02906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000700596; MC1012; NCI-2011-01083; 8810 (Other: Mayo Clinic in Rochester); 8810 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH); NCT02876068 (obsolete NCT alias)
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Melanoma; Refractory Malignant Solid Neoplasm; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Melanoma | interventions — cediranib; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cediranib maleate, selumetinib) (Experimental): Patients receive cediranib maleate PO QD and selumetinib sulfate PO QD or BID on days 1-28 (days 8-28 of cycle 1). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cycles may be extended to 12 weeks after 1 year of study treatment.
  Interventions: Drug: Cediranib; Drug: Cediranib Maleate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Selumetinib; Drug: Selumetinib Sulfate

INTERVENTIONS:
Drug: Cediranib — Given PO
  Other Names: AZ-D2171; AZD 2171; AZD2171
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD 6244; AZD-6244; AZD6244; MEK Inhibitor AZD6244
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate

SUMMARY:
This phase I trial studies the side effects and best dose of cediranib maleate and selumetinib sulfate in treating patients with solid malignancies. Cediranib maleate and selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cediranib maleate may also stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose of cediranib maleate (AZD2171 [cediranib]) in combination with selumetinib sulfate (AZD6244 hydrogen sulfate).

II. To describe the toxicity profile associated with AZD2171 (cediranib) in combination with AZD6244 hydrogen sulfate.

III. To describe the tumor responses and identify any activity of this AZD2171 (cediranib) in combination with AZD6244 hydrogen sulfate.

IV. To explore, through correlative studies, the effect of AZD2171 (cediranib) with or without AZD6244 hydrogen sulfate on serum markers of apoptosis.

V. To assess the pharmacokinetic interaction of AZD2171 (cediranib) in combination with AZD6244 hydrogen sulfate.

VI. To study the association of clinical (toxicity and/or tumor response or activity) with the pharmacologic (pharmacokinetic/pharmacodynamic) parameters, and/or biologic (correlative laboratory study) results.

OUTLINE: This is a dose-escalation study followed by a dose-expansion cohort study.

Patients receive cediranib maleate orally (PO) once daily (QD) and selumetinib sulfate PO QD or twice daily (BID) on days 1-28 (days 8-28 of cycle 1). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cycles may be extended to 12 weeks after 1 year of study treatment.

After completion of study therapy, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now considered clinically unresectable and for whom there is no standard therapy; NOTE: for the maximum tolerated dose (MTD) expansion cohort only: metastatic melanoma histology is required
* Measurable and non-measurable disease are eligible
* Ability to provide informed consent
* Absolute neutrophil count (ANC) >= 1500/uL (obtained =< 21 days prior to registration)
* Platelets (PLT) >= 100,000/uL (obtained =< 21 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 21 days prior to registration)
* Aspartate aminotransferase (AST) =< 2.5 x ULN or =< 5 x ULN in presence of liver metastases (obtained =< 21 days prior to registration)
* Creatinine =< 1.5 x ULN (obtained =< 21 days prior to registration)
* Hemoglobin (HgB) >= 9.0 gm/dL (obtained =< 21 days prior to registration)
* Alkaline phosphatase =< 2.5 x ULN (obtained =< 21 days prior to registration)
* Creatinine clearance > 50 ml/min, by either Cockcroft-Gault formula or 24-hour urine collection analysis (obtained =< 21 days prior to registration)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1
* Willing to return to Mayo for follow up
* Life expectancy >= 12 weeks
* Women of childbearing potential only: negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Expansion phase only: willing to provide blood samples and archived tumor tissue for correlative research purposes

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 28 days prior to registration
  * Mitomycin C/nitrosoureas =< 42 days prior to registration
  * Immunotherapy =< 28 days prior to registration
  * Biologic therapy =< 28 days prior to registration
  * Radiation therapy =< 28 days prior to registration
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* Cardiac conditions as follows:

  * Uncontrolled hypertension (blood pressure [BP] >= 150/95 despite optimal therapy)
  * Heart failure New York Heart Association (NYHA) class II or above or left ventricular ejection fraction < 50%
  * Atrial fibrillation with heart rate > 100 beats per minute (bpm)
  * Unstable ischemic heart disease (myocardial infarction [MI] within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly)
  * Patients who require concomitant agents that prolong corrected QT interval (QTc)
* Known brain or central nervous system (CNS) metastases without definitive therapy; patients who have received definitive therapy for CNS lesions may be considered if there is no evidence of progression on computed tomography (CT) or magnetic resonance imaging (MRI) imaging obtained 3 months apart
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) with the exception of patients known to be human immunodeficiency virus [HIV] positive and have a cluster of differentiation [CD]4 count > 400 and do not require antiretroviral therapy
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment (i.e. hormonal therapy) for their cancer
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart unless urinary protein < 1.5g in a 24 hour (hr) period or urine protein/creatinine ratio < 1.5
* History of exposure to AZD2171 (cediranib), AZD6244 hydrogen sulfate, or mitogen-activated protein kinase kinase (MEK), retrovirus-associated deoxyribonucleic acid (DNA) sequence (Ras) or v-RAF-1 murine leukemia viral oncogene homolog (Raf) inhibitors (sorafenib); Note: prior therapy with bevacizumab, sunitinib, pazopanib or aflibercept (vascular endothelial growth factor [VEGF] Trap) are allowed
* Surgery within two weeks prior to registration
* Significant hemorrhage (> 30 mL bleeding/episode in previous 3 months) or hemoptysis (> 5 mL fresh blood in previous 4 weeks)
* Mean QTc interval with Bazetts correction > 480 msec (Common Toxicity Criteria [CTC] grade 1) in screening electrocardiogram (ECG) or history of familial long QT syndrome
* Patients who are unable to swallow tablets and capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days
  MTD will be defined as the dose level below the lowest dose that induces dose limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients). Graded per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).

SECONDARY OUTCOMES:
Incidence of adverse events, classified as either possibly, probably, or definitely related to study treatment | Up to 3 months
  Will be assessed using NCI CTCAE. The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Incidence of hematologic toxicities | Up to 3 months
  Will be evaluated via Common Toxicity Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization.
Incidence of non-hematologic toxicities | Up to 3 months
  Will be evaluated via the ordinal CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Overall toxicity incidence | Up to 3 months
  Will be evaluated using NCI CTCAE. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Best response | From the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started), assessed up to 3 months
  Will be evaluated using Response Evaluation Criteria in Solid Tumors 1.1 criteria. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).

OTHER OUTCOMES:
Changes of the serum levels of M30 (dose expansion phase) | Baseline up to day 22 of course 1
  Descriptive statistics, scatter plots and longitudinal data plot will form the basis of presentation of these data. Multiple comparison corrections (e.g. Bonferroni) will be performed during data analyses.
Changes of the serum levels of caspase 3 (dose expansion phase) | Baseline up to day 22 of course 1
  Descriptive statistics, scatter plots and longitudinal data plot will form the basis of presentation of these data. Multiple comparison corrections (e.g. Bonferroni) will be performed during data analyses.
Changes of the serum levels of cytochrome c (dose expansion phase) | Baseline up to day 22 of course 1
  Descriptive statistics, scatter plots and longitudinal data plot will form the basis of presentation of these data. Multiple comparison corrections (e.g. Bonferroni) will be performed during data analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Costello, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Emiloju OE, Yin J, Koubek E, Reid JM, Borad MJ, Lou Y, Seetharam M, Edelman MJ, Sausville EA, Jiang Y, Kaseb AO, Posey JA, Davis SL, Gores GJ, Roberts LR, Takebe N, Schwartz GK, Hendrickson AEW, Kaufmann SH, Adjei AA, Hubbard JM, Costello BA. Phase 1 trial of navitoclax and sorafenib in patients with relapsed or refractory solid tumors with hepatocellular carcinoma expansion cohort. Invest New Drugs. 2024 Feb;42(1):127-135. doi: 10.1007/s10637-024-01420-8. Epub 2024 Jan 25. PMID 38270822